CLINICAL TRIAL: NCT02690454
Title: Which Platelet Function Test Provides the Best Reflection of the in Vivo Plasma Concentrations of Ticagrelor and Its Active Metabolite? A Pharmacokinetic and Pharmacodynamic Study Including Patients With Myocardial Infarction.
Brief Title: Which Platelet Function Test Best Reflects the In Vivo Plasma Concentrations of Ticagrelor and Its Active Metabolite?
Acronym: HARMONIC
Status: Completed | Type: Observational
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Marek Kozinski, Principal Investigator, Assoc. Prof., MD, PhD, FESC, Collegium Medicum w Bydgoszczy
Other Study IDs: CMUMK202E
Record Dates: First submitted 2015-11-26; First posted 2016-02-24 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Infarction; Myocardial Infarction; Cardiovascular Diseases; Heart Diseases; Ischemia; Myocardial Ischemia; Necrosis; Pathologic Processes; Vascular Diseases
Keywords: ticagrelor; ticagrelor active metabolite (AR-C124910XX); platelet function tests; the flow cytometric VASP assay; the VerifyNow® device; the Multiplate® analyzer; pharmacokinetics; pharmacodynamics; Multiplate® ADPtest; VerifyNow® PRUTest™; Platelet VASP/P2Y12 assay
MeSH Terms: conditions — Infarction; Myocardial Infarction; Cardiovascular Diseases; Heart Diseases; Ischemia; Myocardial Ischemia; Necrosis; Pathologic Processes; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ticagrelor is a direct-acting, reversible platelet P2Y12 receptor inhibitor recommended by the recent European Society of Cardiology guidelines in patients with acute coronary syndromes (ACS) (class of recommendation I, level of evidence B). Ticagrelor inhibits platelet function stronger, faster and more consistently than clopidogrel, the former standard of antiplatelet therapy. In the landmark PLATO trial (Study of PLATelet inhibition and patient Outcomes), ticagrelor therapy as compared with clopidogrel treatment was associated with the reduced occurrence of major adverse cardiovascular events and all-cause mortality, but also resulted in a small, but statistically significant, increase in the rate of major bleeding. The optimum choice of antiplatelet treatment, aimed to provide each patient with maximum protection against ischemic events, while minimizing the risk of bleeding complications, is the challenge of contemporary ACS therapy. The tool which may help physicians and facilitate clinical decision making is platelet function testing. According to the guidance of both European and American groups of experts, there are three currently recommended platelet function tests, namely the VerifyNow device, the Multiplate analyzer and the Vasodilator Stimulated Phosphoprotein Phosphorylation (VASP) assay. It needs to be emphasized that none of these three methods is preferred over others. So far there are no studies linking pharmacokinetic analysis of ticagrelor and its active metabolite with comparative evaluation of platelet reactivity. The aim of this trial is to assess the relationship between concentrations of ticagrelor and its active metabolite (AR-C124910XX) and results of all three recommended platelet function tests in patients with myocardial infarction. Patients who receive GP IIb/IIIa receptor inhibitor will be excluded from the primary analysis.

Statistical analysis: The correlation will be assessed using correlation coefficients and intraclass correlation coefficients. while the agreement between the results of the compared platelet function tests will be measured using the Kappa statistic and Bland-Altman analysis.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent prior to any study specific procedures
* diagnosis of acute ST-segment elevation myocardial infarction or acute non-ST-segment
* male or non-pregnant female, aged 18-80 years old
* provision of informed consent for angiography and PCI

Exclusion Criteria:

* treatment with ticlopidine, clopidogrel, prasugrel or ticagrelor within 14 days before the study enrollment
* hypersensitivity to ticagrelor
* current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* active bleeding
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of coagulation disorders
* platelet count less than <100 x10^3/mcl
* hemoglobin concentration less than 10.0 g/dl
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* patients considered by the investigator to be at risk of bradycardic events
* second or third degree atrioventricular block during screening for eligibility
* history of asthma or severe chronic obstructive pulmonary disease
* patient required dialysis
* manifest infection or inflammatory state
* Killip class III or IV during screening for eligibility
* respiratory failure
* history of severe chronic heart failure (NYHA class III or IV)
* concomitant therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir) or strong CYP3A inducers (rifampicin, phenytoin, carbamazepine, dexamethasone, phenobarbital) within 14 days and during study treatment
* body weight below 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myocardial infarction
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between ticagrelor plasma concentration and platelet reactivity measurement [platelet reactivity index (PRI), platelet arbitrary aggregation units/min and P2Y12 Reaction Units (PRU)]. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess correlation coefficients in broad ranges of ticagrelor concentrations and values of platelet reactivity. Platelet reactivity measurements will be made immediately after blood sample collection. Ticagrelor plasma concentration will be assessed at the end of participant enrollment. From each study participant, 8 correlation coefficients (for eight sampling points) for each compared methods of platelet reactivity measurement will be included in the final analysis. Values of correlation coefficients will be compared among assessed methods of platelet reactivity measurement.
  Platelet reactivity measurements: platelet reactivity index (PRI) assessed by VASP/P2Y12 assay, platelet arbitrary aggregation units/min assessed by Multiple Electrode Aggregometry (Multiplate® ADPtest) and P2Y12 Reaction Units (PRU) assessed by VerifyNow® PRUTest™.

SECONDARY OUTCOMES:
Correlation coefficient between ticagrelor active metabolite (AR-C124910XX) plasma concentration and platelet reactivity measurement [platelet reactivity index (PRI), platelet arbitrary aggregation units/min and P2Y12 Reaction Units (PRU)]. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess correlation coefficients in broad ranges of AR-C124910XX concentrations and values of platelet reactivity. Platelet reactivity measurements will be made immediately after blood sample collection. Active ticagrelor metabolite plasma concentration will be assessed at the end of participant enrollment. From each study participant, 8 correlation coefficients (for eight sampling points) for each compared methods of platelet reactivity measurement will be included in the final analysis. Values of correlation coefficients will be compared among assessed methods of platelet reactivity measurement at the end of participant enrollment.
  Platelet reactivity measurements: platelet reactivity index (PRI) assessed by VASP/P2Y12 assay, platelet arbitrary aggregation units/min assessed by Multiple Electrode Aggregometry (Multiplate® ADPtest) and P2Y12 Reaction Units (PRU) assessed by VerifyNow® PRUTest™.
Correlation coefficient between ticagrelor plasma concentration and inhibition of platelet reactivity assessed with VASP assay, Multiplate® analyzer and VerifyNow® device). | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess correlation coefficients in broad ranges of ticagrelor concentrations and values of inhibition of platelet reactivity. From each study participant, 7 correlation coefficients (for inhibition of platelet reactivity 1, 2, 3, 4, 6, 12, 24 hours post dose) for each compared methods of platelet reactivity measurement will be included in the final analysis. Values of correlation coefficients will be calculated and compared among assessed methods of platelet reactivity measurement at the end of participant enrollment.
  Inhibition of platelet aggregation: predose platelet reactivity minus actual platelet reactivity divided by predose platelet reactivity.
  Platelet reactivity measurements: platelet reactivity index (PRI) assessed by VASP/P2Y12 assay, platelet arbitrary aggregation units/min assessed by Multiple Electrode Aggregometry (Multiplate® ADPtest) and P2Y12 Reaction Units (PRU) assessed by VerifyNow® PRUTest™.
Correlation coefficient between ticagrelor active metabolite (AR-C124910XX) plasma concentration and inhibition of platelet reactivity assessed with VASP assay, Multiplate® analyzer and VerifyNow® device. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess correlation coefficients in broad ranges of AR-C124910XX concentrations and values of inhibition of platelet reactivity. From each study participant, 7 correlation coefficients (for inhibition of platelet reactivity 1, 2, 3, 4, 6, 12, 24 hours post dose) for each compared methods of platelet reactivity measurement will be included in the final analysis. Values of correlation coefficients will be calculated and compared among assessed methods of platelet reactivity measurement at the end of participant enrollment.
  Inhibition of platelet aggregation: predose platelet reactivity minus actual platelet reactivity divided by predose platelet reactivity.
  Platelet reactivity measurements: platelet reactivity index (PRI) assessed by VASP/P2Y12 assay, platelet arbitrary aggregation units/min assessed by Multiple Electrode Aggregometry (Multiplate® ADPtest) and P2Y12 Reaction Units (PRU) assessed by VerifyNow® PRUTest™.
Kappa statistics assessing agreement between the platelet reactivity measurements performed with the VASP assay and the Multiplate® and VerifyNow® assays in terms of identification of patients with high on-ticagrelor platelet reactivity. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess a broad range of platelet reactivity values. From each study participant, eight measurements of platelet reactivity (for all sampling points) for each compared methods will be included in the final analysis.The Kappa statistics values will be calculated at the end of participant enrollment.
Kappa statistics assessing agreement between the platelet reactivity measurements performed with the Multiplate® assay and the VASP and VerifyNow® assays in terms of identification of patients with low on-ticagrelor platelet reactivity. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected collected in multiple time points in order to assess a broad range of platelet reactivity values. From each study participant, eight measurements of platelet reactivity (for all sampling points) for each compared methods will be included in the final analysis.The Kappa statistics values will be calculated at the end of participant enrollment.
Correlation coefficient between the standardized values of platelet reactivity performed with the Multiplate® assay and the VASP and VerifyNow® assays. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess a broad range of platelet reactivity values. From each study participant, eight measurements of platelet reactivity (for all sampling points) for each compared methods will be included in the final analysis. Values of correlation coefficients will be calculated and compared among assessed methods of platelet reactivity measurement at the end of participant enrollment.
  Standardized platelet reactivity: actual platelet reactivity minus mean platelet reactivity divided by standardized deviation of the platelet reactivity.
Intraclass correlation coefficient between the standardized values of platelet reactivity performed with the Multiplate® assay and the VASP and VerifyNow® assays. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess a broad range of platelet reactivity values. From each study participant, eight measurements of platelet reactivity (for all sampling points) for each compared methods will be included in the final analysis. Values of intraclass correlation coefficients will be calculated and compared among assessed methods of platelet reactivity measurement at the end of participant enrollment.
  Standardized platelet reactivity: actual platelet reactivity minus mean platelet reactivity divided by standardized deviation of the platelet reactivity.
Blant-Altman analysis assessing agreement between the standardized values of platelet reactivity performed with the Multiplate® assay and the VASP and VerifyNow® assays. | predose, 1, 2, 3, 4, 6, 12, 24 hours post-dose
  Blood samples will be collected in multiple time points in order to assess a broad range of platelet reactivity values. From each study participant, eight measurements of platelet reactivity (for all sampling points) for each compared methods will be included in the final analysis. Bland-Altman analysis will be performed at the end of participant enrollment.
  Standardized platelet reactivity: actual platelet reactivity minus mean platelet reactivity divided by standardized deviation of the platelet reactivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland